CLINICAL TRIAL: NCT06204276
Title: The Physiologic Effects of Asymmetrical Versus Conventional High-flow Nasal Cannula in Acute Respiratory Failure. A Randomized Crossover Study.
Brief Title: Asymmetrical Versus Conventional High-flow Nasal Cannula in Acute Respiratory Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Nuttapol Rittayamai, Associate Professor, Siriraj Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 763/2566(IRB4)
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Acute Hypoxemic Respiratory Failure; Acute Hypercapnic Respiratory Failure
Keywords: high-flow nasal cannula; respiratory failure; respiratory muscles; ultrasound
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Asymmetrical high-flow nasal cannula (Experimental): * Asymmetrical nasal cannula (Optiflow+ Duet nasal cannula)
  * Airvo-2 (Fisher&Paykel)
  Interventions: Device: Experimental: Asymmetrical high-flow nasal cannula
- Conventional high-flow nasal cannula (Active Comparator): * Conventional nasal cannula (Optiflow+ nasal cannula)
  * Airvo-2 (Fisher&Paykel)
  Interventions: Device: Active comparator: Conventional high-flow nasal cannula

INTERVENTIONS:
Device: Experimental: Asymmetrical high-flow nasal cannula — Asymmetrical high-flow nasal cannula will be set at 40 and 60 L/min in a random order. Temperature will be set at 37 degree celsius and inspired oxygen fraction (FiO2) will be adjusted to maintain oxygen saturation by pulse oximetry (SpO2) >/= 94% in acute hypoxemic patients and between 92-94% in acute hypercapnic COPD patients
  Arms: Asymmetrical high-flow nasal cannula
Device: Active comparator: Conventional high-flow nasal cannula — Conventional high-flow nasal cannula will be set at 40 and 60 L/min in a random order. Temperature will be set at 37 degree celsius and FiO2 will be adjusted to maintain SpO2 >/= 94% in acute hypoxemic patients and between 92-94% in acute hypercapnic COPD patients
  Arms: Conventional high-flow nasal cannula

SUMMARY:
The goal of this randomized crossover physiological study is to evaluate the physiologic effects of asymmetrical nasal cannula and conventional nasal cannula in patients with acute respiratory failure. The main questions it aims to answer are:

* Does the asymmetrical high-flow nasal cannula reduce the diaphragm and parasternal intercostal work activity of breathing measured by ultrasound compared to conventional high-flow nasal cannula?
* What is the effect of the asymmetrical high-flow nasal cannula on breathing pattern, gas exchange, and hemodynamic variables compared to conventional high-flow nasal cannula? Participants will received asymmetrical high-flow nasal cannula or conventional high-flow nasal cannula at a flow rate of 40 and 60 L/min in a random order.

DETAILED DESCRIPTION:
High-flow nasal cannula (HFNC) is increasingly used in patients with acute respiratory failure. The physiologic benefits of HFNC can be explained via several mechanisms. These mechanisms lead to improve alveolar ventilation and decrease patient's inspiratory effort directly or indirectly.

Recent clinical practice guidelines recommended to use HFNC in patients with acute hypoxemic respiratory failure over conventional oxygen therapy (COT) and noninvasive ventilation (NIV). A landmark clinical study demonstrated that patients with acute hypoxemic respiratory failure who received HFNC had better survival than COT and NIV. A systematic review and meta-analysis also demonstrated that HFNC significantly reduced escalation of respiratory support in patients with acute hypoxemic respiratory failure.

HFNC can also be an alternative respiratory support in patients with acute on chronic hypercapnic chronic obstructive pulmonary disease (COPD). Several physiological and clinical studies in COPD patients with exacerbations have also suggested that HFNC was not inferior to noninvasive ventilation (NIV) in COPD patients with mild to moderate exacerbation, in terms of gas exchange, treatment failure, intubation rate, and mortality rate. It may be also be used during NIV interruptions or after extubation.

Recently, an asymmetrical HFNC interface has been developed with a feature of one prong of smaller diameter and the other prong of larger diameter resulting in an increase in the overall cross-sectional area compared to conventional HFNC interface. An experimental study has shown that asymmetrical nasal cannula potentially increased positive end-expiratory pressure (PEEP) and enhanced carbon dioxide washout compared to conventional nasal cannula. Different respective effects in terms of pressure, resistance, and dead space washout between the two types of cannulas may explain different results, according to the population.

The aim of this study is to evaluate the physiologic effects of asymmetrical nasal cannula and conventional nasal cannula on diaphragm and parasternal intercostal activity of breathing measured by ultrasound in patients with acute respiratory failure.

ELIGIBILITY:
Patients with acute hypoxemia respiratory failure

Inclusion Criteria:

* Age > 18 years old
* Acute respiratory failure within 7 days of hospital admission?
* Hypoxemia defined by arterial partial pressure of oxygen (PaO2)/FiO2 < 300 mmHg or SpO2/FiO2 < 315
* Already supported with HFNC device

Exclusion Criteria:

* Respiratory acidosis: pH < 7.30 and PaCO2 > 45 mmHg
* Hemodynamic instability requiring vasopressor initiation
* Diminished level of consciousness or uncooperative
* Active hemoptysis or pneumothorax requiring a chest tube
* Chronic severe neuromuscular disease
* Pregnancy

Patients with acute hypercapnic COPD Inclusion criteria

* Age > 40 years old
* Diagnosed COPD according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) guideline (postbronchodilator forced expiratory volume at 1 second (FEV1)/forced vital capacity (FVC) < 70%)
* Exacerbation requiring hospitalization; at least 2 of the following criteria

  1. Respiratory rate > 24/min
  2. Use of respiratory accessory muscles or paradoxical motion of the abdomen
  3. Acute respiratory acidosis with arterial or venous pH < 7.35 and/or PaCO2 > 45 mmHg

Exclusion criteria

* pH < 7.25
* Hemodynamic instability requiring vasopressor initiation
* Persistent hypoxemia despite supplemental oxygen therapy
* Diminished level of consciousness or uncooperative
* Active hemoptysis or pneumothorax requiring a chest tube
* Associated severe chronic neuromuscular disease
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Diaphragm thickening fraction | 15 minutes
  Diaphragm thickening fraction measured by ultrasound

SECONDARY OUTCOMES:
Parasternal intercostal thickening fraction | 15 minutes
  Parasternal intercostal thickening fraction measured by ultrasound
Parasternal intercostal/diaphragm thickening fraction ratio | 15 minutes
  Contribution between parasternal intercostal and diaphragm thickening fraction
Respiratory rate | 15 minutes
  Respiratory rate
Oxygen saturation | 15 minutes
  Pulse oximetry
Transcutaneous carbon dioxide (CO2) pressure | 15 minutes
  Transcutaneous CO2 monitor
Mean arterial pressure | 15 minutes
  Blood pressure
Heart rate | 15 minutes
  Heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Nuttapol Rittayamai, M.D., Principal Investigator — Siriraj Hospital
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ricard JD, Roca O, Lemiale V, Corley A, Braunlich J, Jones P, Kang BJ, Lellouche F, Nava S, Rittayamai N, Spoletini G, Jaber S, Hernandez G. Use of nasal high flow oxygen during acute respiratory failure. Intensive Care Med. 2020 Dec;46(12):2238-2247. doi: 10.1007/s00134-020-06228-7. Epub 2020 Sep 8. PMID 32901374
- [Background] Biselli P, Fricke K, Grote L, Braun AT, Kirkness J, Smith P, Schwartz A, Schneider H. Reductions in dead space ventilation with nasal high flow depend on physiological dead space volume: metabolic hood measurements during sleep in patients with COPD and controls. Eur Respir J. 2018 May 30;51(5):1702251. doi: 10.1183/13993003.02251-2017. Print 2018 May. PMID 29724917
- [Background] Vieira F, Bezerra FS, Coudroy R, Schreiber A, Telias I, Dubo S, Cavalot G, Pereira SM, Piraino T, Brochard LJ. High Flow Nasal Cannula compared to Continuous Positive Airway Pressure: a bench and physiological study. J Appl Physiol (1985). 2022 May 5. doi: 10.1152/japplphysiol.00416.2021. Online ahead of print. PMID 35511720
- [Background] Mauri T, Turrini C, Eronia N, Grasselli G, Volta CA, Bellani G, Pesenti A. Physiologic Effects of High-Flow Nasal Cannula in Acute Hypoxemic Respiratory Failure. Am J Respir Crit Care Med. 2017 May 1;195(9):1207-1215. doi: 10.1164/rccm.201605-0916OC. PMID 27997805
- [Background] Rittayamai N, Phuangchoei P, Tscheikuna J, Praphruetkit N, Brochard L. Effects of high-flow nasal cannula and non-invasive ventilation on inspiratory effort in hypercapnic patients with chronic obstructive pulmonary disease: a preliminary study. Ann Intensive Care. 2019 Oct 22;9(1):122. doi: 10.1186/s13613-019-0597-5. PMID 31641959
- [Background] Rochwerg B, Einav S, Chaudhuri D, Mancebo J, Mauri T, Helviz Y, Goligher EC, Jaber S, Ricard JD, Rittayamai N, Roca O, Antonelli M, Maggiore SM, Demoule A, Hodgson CL, Mercat A, Wilcox ME, Granton D, Wang D, Azoulay E, Ouanes-Besbes L, Cinnella G, Rauseo M, Carvalho C, Dessap-Mekontso A, Fraser J, Frat JP, Gomersall C, Grasselli G, Hernandez G, Jog S, Pesenti A, Riviello ED, Slutsky AS, Stapleton RD, Talmor D, Thille AW, Brochard L, Burns KEA. The role for high flow nasal cannula as a respiratory support strategy in adults: a clinical practice guideline. Intensive Care Med. 2020 Dec;46(12):2226-2237. doi: 10.1007/s00134-020-06312-y. Epub 2020 Nov 17. PMID 33201321
- [Background] Nagata K, Horie T, Chohnabayashi N, Jinta T, Tsugitomi R, Shiraki A, Tokioka F, Kadowaki T, Watanabe A, Fukui M, Kitajima T, Sato S, Tsuda T, Kishimoto N, Kita H, Mori Y, Nakayama M, Takahashi K, Tsuboi T, Yoshida M, Hataji O, Fuke S, Kagajo M, Nishine H, Kobayashi H, Nakamura H, Okuda M, Tachibana S, Takata S, Osoreda H, Minami K, Nishimura T, Ishida T, Terada J, Takeuchi N, Kohashi Y, Inoue H, Nakagawa Y, Kikuchi T, Tomii K. Home High-Flow Nasal Cannula Oxygen Therapy for Stable Hypercapnic COPD: A Randomized Clinical Trial. Am J Respir Crit Care Med. 2022 Dec 1;206(11):1326-1335. doi: 10.1164/rccm.202201-0199OC. PMID 35771533
- [Background] Cortegiani A, Longhini F, Madotto F, Groff P, Scala R, Crimi C, Carlucci A, Bruni A, Garofalo E, Raineri SM, Tonelli R, Comellini V, Lupia E, Vetrugno L, Clini E, Giarratano A, Nava S, Navalesi P, Gregoretti C; H. F.-AECOPD study investigators. High flow nasal therapy versus noninvasive ventilation as initial ventilatory strategy in COPD exacerbation: a multicenter non-inferiority randomized trial. Crit Care. 2020 Dec 14;24(1):692. doi: 10.1186/s13054-020-03409-0. PMID 33317579
- [Background] Lee MK, Choi J, Park B, Kim B, Lee SJ, Kim SH, Yong SJ, Choi EH, Lee WY. High flow nasal cannulae oxygen therapy in acute-moderate hypercapnic respiratory failure. Clin Respir J. 2018 Jun;12(6):2046-2056. doi: 10.1111/crj.12772. Epub 2018 Mar 5. PMID 29392846
- [Background] Longhini F, Pisani L, Lungu R, Comellini V, Bruni A, Garofalo E, Laura Vega M, Cammarota G, Nava S, Navalesi P. High-Flow Oxygen Therapy After Noninvasive Ventilation Interruption in Patients Recovering From Hypercapnic Acute Respiratory Failure: A Physiological Crossover Trial. Crit Care Med. 2019 Jun;47(6):e506-e511. doi: 10.1097/CCM.0000000000003740. PMID 30882477
- [Background] Tan D, Walline JH, Ling B, Xu Y, Sun J, Wang B, Shan X, Wang Y, Cao P, Zhu Q, Geng P, Xu J. High-flow nasal cannula oxygen therapy versus non-invasive ventilation for chronic obstructive pulmonary disease patients after extubation: a multicenter, randomized controlled trial. Crit Care. 2020 Aug 6;24(1):489. doi: 10.1186/s13054-020-03214-9. PMID 32762701
- [Background] Tatkov S, Rees M, Gulley A, van den Heuij LGT, Nilius G. Asymmetrical nasal high flow ventilation improves clearance of CO2 from the anatomical dead space and increases positive airway pressure. J Appl Physiol (1985). 2023 Feb 1;134(2):365-377. doi: 10.1152/japplphysiol.00692.2022. Epub 2023 Jan 12. PMID 36633864
- [Background] Slobod D, Spinelli E, Crotti S, Lissoni A, Galazzi A, Grasselli G, Mauri T. Effects of an asymmetrical high flow nasal cannula interface in hypoxemic patients. Crit Care. 2023 Apr 18;27(1):145. doi: 10.1186/s13054-023-04441-6. PMID 37072854
- [Background] Goligher EC, Laghi F, Detsky ME, Farias P, Murray A, Brace D, Brochard LJ, Bolz SS, Rubenfeld GD, Kavanagh BP, Ferguson ND. Measuring diaphragm thickness with ultrasound in mechanically ventilated patients: feasibility, reproducibility and validity. Intensive Care Med. 2015 Apr;41(4):642-9. doi: 10.1007/s00134-015-3687-3. Epub 2015 Feb 19. PMID 25693448
- [Background] Zambon M, Greco M, Bocchino S, Cabrini L, Beccaria PF, Zangrillo A. Assessment of diaphragmatic dysfunction in the critically ill patient with ultrasound: a systematic review. Intensive Care Med. 2017 Jan;43(1):29-38. doi: 10.1007/s00134-016-4524-z. Epub 2016 Sep 12. PMID 27620292
- [Background] Vivier E, Mekontso Dessap A, Dimassi S, Vargas F, Lyazidi A, Thille AW, Brochard L. Diaphragm ultrasonography to estimate the work of breathing during non-invasive ventilation. Intensive Care Med. 2012 May;38(5):796-803. doi: 10.1007/s00134-012-2547-7. Epub 2012 Apr 5. PMID 22476448